CLINICAL TRIAL: NCT02806960
Title: A Single Center, Randomized, 4-Period Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Single or Repeated 3 mg Doses of Intranasally Administered Glucagon in Adults With Type 1 or Type 2 Diabetes
Brief Title: A Study of Single and Repeated Doses of Glucagon Administered to Participants With Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug delivery was below target dose due to partial obstruction by aggregated particles.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16493; I8R-MC-IGBH (Other: Eli Lilly and Company); AMG110 (Other: AMG Medical Inc); AMG-P4-459 (Other: AMG Medical Inc)
Record Dates: First submitted 2016-05-26; First posted 2016-06-21 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (Experimental): Treatment 1, single nasal glucagon (NG) dose of 3 milligram (mg).
  Interventions: Drug: Nasal Glucagon
- Treatment 2 (Experimental): Treatment 2, NG dose of 3 mg plus 3 mg NG dose in same nostril 15 minutes later.
  Interventions: Drug: Nasal Glucagon
- Treatment 3 (Experimental): Treatment 3, NG dose of 3 mg plus 3 mg NG dose in the opposite nostril 15 minutes later.
  Interventions: Drug: Nasal Glucagon
- Treatment 4 (Experimental): Treatment 4, NG dose of 3 mg then immediately 3 mg NG dose in the opposite nostril.
  Interventions: Drug: Nasal Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon — Administered intranasally.
  Other Names: LY900018; AMG 504-1

SUMMARY:
This study will investigate how the body processes nasal glucagon and the effect of nasal glucagon on the body. After an 8-hour overnight fast and 4 hours after the start of a low-carbohydrate breakfast, the study drug will be delivered into the participant's nostril(s) (intranasally) once or twice in each of four study periods. The study is open to adults with type 1 or type 2 diabetes and is expected to last about 50 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with a history of Type 1 or Type 2 insulin-using diabetes of at least 1 year duration (basal only, basal bolus, meal-time only, or twice a day pre-mixed insulin)
* A female participant must meet one of the following criteria:

  * Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first administration of the study drug, during the study and for at least 30 days after the last dose of the study drug.
  * Participant is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses)
* Participants with a body mass index (BMI) greater than or equal to 18.50 kilograms per square meter (kg/m²) and below 35.00 kg/m²
* Light-, non- or ex-smokers
* In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the Investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations

Exclusion Criteria:

* Females who are pregnant, actively attempting to get pregnant, or are lactating
* History of significant hypersensitivity to glucagon or any related products as well as severe hypersensitivity reactions (such as angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions which in the judgment of the Investigator could interfere with the absorption, distribution, metabolism or excretion of drugs, or could potentiate or predispose to undesired effects
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Known presence of rare hereditary problems of galactose and /or lactose intolerance
* Known presence or history of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma (i.e. insulin secreting pancreas tumor) Presence of clinically significant findings on nasal examination or bilateral anterior rhinoscopy, such as structural abnormalities, nasal polyps, marked septal deviation, nasal tumors
* Nasal surgery in the previous 28 days before Day 1 of this study
* Daily use of a systemic beta-blocker drug, indomethacin, warfarin or anticholinergic drugs in the previous 28 days before Day 1 of this study
* Any other concomitant maintenance therapy that would influence the outcome of the trial or compromise the safety of the participant, at the discretion of the Investigator and the Sponsor, in the previous 28 days before Day 1 of this study
* Significant history of drug dependency or alcohol abuse
* Any clinically significant illness in the previous 28 days before Day 1 of this study
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive urine screening of alcohol and/or drugs of abuse
* Concurrent participation or intention of participating in another clinical trial during this study
* Participants who took an Investigational Product (in another clinical trial) in the previous 28 days before Day 1 of this study or who have already participated in this clinical study
* Participants who donated 50 milliliters (mL) or more of blood in the previous 28 days before Day 1 of this study
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before Day 1 of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4-period, 4 sequence, repeated single dose design with 7 days washout period between each dose.
Groups:
- Sequence 1 (Treatment 1, 2, 3 and 4): The intranasal (IN) glucagon formulation was randomly administered in the morning after a 8-hour overnight fast and 4 hours after the start of a low-carbohydrate breakfast, as per below sequence:
  Period 1: Single 3 mg dose of Nasal glucagon (NG).
  Period 2: Single 3 mg dose of Nasal Glucagon at time 0, followed by a second 3 mg dose of Nasal Glucagon 15 minutes later in the same nostril (for a total of 6 mg of glucagon).
  Period 3: Single 3 mg dose of Nasal Glucagon at time 0, followed by a second 3 mg dose of Nasal Glucagon 15 minutes later in the opposite nostril (for a total of 6 mg of glucagon).
  Period 4: Single 3 mg dose of Nasal Glucagon at time 0, followed by a second 3 mg dose of Nasal Glucagon immediately after (within 1 minute) in the opposite nostril (for a total of 6 mg of glucagon).
- Sequence 2 (Treatment 2, 3, 4 and 1): The Intranasal glucagon formulation was randomly administered in the morning after a 8-hour overnight fast and 4 hours after the start of a low-carbohydrate breakfast, as per below sequence:
  Period 1: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG 15 minutes later in the same nostril (for a total of 6 mg of glucagon).
  Period 2: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG 15 minutes later in the opposite nostril (for a total of 6 mg of glucagon).
  Period 3: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG immediately after (within 1 minute) in the opposite nostril (for a total of 6 mg of glucagon).
  Period 4: Single 3 mg dose of NG.
- Sequence 3 (Treatment 3, 4, 1 and 2): The IN glucagon formulation was randomly administered in the morning after a 8-hour overnight fast and 4 hours after the start of a low-carbohydrate breakfast, as per below sequence:
  Period 1: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG 15 minutes later in the opposite nostril (for a total of 6 mg of glucagon).
  Period 2: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG immediately after (within 1 minute) in the opposite nostril (for a total of 6 mg of glucagon).
  Period 3: Single 3 mg dose of NG.
  Period 4: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG 15 minutes later in the same nostril (for a total of 6 mg of glucagon).
- Sequence 4 (Treatment 4, 1, 2 and 3): The IN glucagon formulation was randomly administered in the morning after a 8-hour overnight fast and 4 hours after the start of a low-carbohydrate breakfast, as per below sequence:
  Period 1: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG immediately after (within 1 minute) in the opposite nostril (for a total of 6 mg of glucagon).
  Period 2: Single 3 mg dose of NG.
  Period 3: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG 15 minutes later in the same nostril (for a total of 6 mg of glucagon).
  Period 4: Single 3 mg dose of NG at time 0, followed by a second 3 mg dose of NG 15 minutes later in the opposite nostril (for a total of 6 mg of glucagon).
Period: Period 1
Arm/Group | Sequence 1 (Treatment 1, 2, 3 and 4) | Sequence 2 (Treatment 2, 3, 4 and 1) | Sequence 3 (Treatment 3, 4, 1 and 2) | Sequence 4 (Treatment 4, 1, 2 and 3)
Started | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3
Not completed — Study Terminated (withdrawn by sponsor) | 3 | 3 | 3 | 3
Period: Period 2
Arm/Group | Sequence 1 (Treatment 1, 2, 3 and 4) | Sequence 2 (Treatment 2, 3, 4 and 1) | Sequence 3 (Treatment 3, 4, 1 and 2) | Sequence 4 (Treatment 4, 1, 2 and 3)
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 (Treatment 1, 2, 3 and 4) | Sequence 2 (Treatment 2, 3, 4 and 1) | Sequence 3 (Treatment 3, 4, 1 and 2) | Sequence 4 (Treatment 4, 1, 2 and 3)
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 (Treatment 1, 2, 3 and 4) | Sequence 2 (Treatment 2, 3, 4 and 1) | Sequence 3 (Treatment 3, 4, 1 and 2) | Sequence 4 (Treatment 4, 1, 2 and 3)
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Participants: A minimum dose of 3 mg NG was administered.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 12

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to T (AUC[0-tlast]) of Baseline Adjusted Glucagon
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.33, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2, 2.5, and 3 hours post dose for each treatment
Population: Zero participants analyzed due to the limited number of samples and the delivery of a potential sub-target dosing dose.
Groups:
- Treatment 1: Single NG dose of 3 mg
- Treatment 2: NG dose of 3 mg plus 3 mg NG dose in same nostril 15 minutes later
- Treatment 3: NG dose of 3 mg plus 3 mg NG dose in the opposite nostril 15 minutes later
- Treatment 4: NG dose of 3 mg then immediately 3 mg NG dose in the opposite nostril.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: PK: Area Under the Curve Extrapolated to Infinity (AUC[0-inf]) of Baseline Adjusted Glucagon
Time Frame: as for outcome 1
Population: Zero participants analyzed due to the limited number of samples and the delivery of a potential sub-target dosing dose.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: PK: Time to Maximum Concentration (Tmax) of Baseline Adjusted Glucagon
Time Frame: as for outcome 1
Population: Zero participants analyzed due to the limited number of samples and the delivery of a potential sub-target dosing dose.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: PK: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: as for outcome 1
Population: Zero participants analyzed due to the limited number of samples and the delivery of a potential sub-target dosing dose.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Pharmacodynamics (PD): Area Under the Effect Concentration Time Curve (AUEC₀-₁.₅) of Blood Glucose (BG)
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.33, 0.5, 0.75, 1.0, 1.25, and 1.5 hours post dose for each treatment
Population: Zero participants analyzed due to the limited number of samples and the delivery of a potential sub-target dosing dose.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: PD: Time to Maximum Concentration (Tmax) of Baseline-Adjusted Glucose
Time Frame: as for outcome 1
Population: Zero participants analyzed due to the limited number of samples and the delivery of a potential sub-target dosing dose.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Primary Outcome: PD: Baseline-Adjusted Glucose Maximum Concentration (BGmax)
Time Frame: as for outcome 1
Population: Zero participants analyzed due to the limited number of samples and the delivery of a potential sub-target dosing dose.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) until study discontinuation (Day 10)
Description: All enrolled participants.
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 (N=3) | Treatment 2 (N=3) | Treatment 3 (N=3) | Treatment 4 (N=3)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Parosmia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study drug was discovered to be delivering a potential sub-target dosing to some participants, due to partial obstruction of the delivery device by aggregation of particles. The study was terminated early with no safety concern for participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days